CLINICAL TRIAL: NCT02001454
Title: Quality of Pain Management at the Ziv Medical Center
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, David Eliya Rothem, Orthopedic Joint Specialist, Ziv Hospital
Other Study IDs: 0032-13
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Focus of the Study Includes Patients in Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients in pain: There is no intervention, only questionnaires for the patient
- Attending Physicians and Nurses: The staff physicians and nurses will also fill out a questionnaire

SUMMARY:
The purpose of this study is to compare attitudes and knowledge of the staff of various departments in our Medical Center in regards to pain treatment. With the results of our survey we will then draw up a protocol on pain management.

DETAILED DESCRIPTION:
Our belief is that the establishment of a pain protocol at the Ziv Medical Center will improve effectiveness of pain treatment. The present study involves surveying the current knowledge and attitudes of caregivers who are responsible for evaluating pain in patients and subsequent treatment in various departments of the hospital without a pain protocol.

According to the IASP (International Association for the Study of Pain) :" Pain is an unpleasant sensory and emotional experience associated with actual or potential tissue damage, or described in terms of such damage". According to WHO, assessment is necessary in every situation that involves pain, excluding pain that is life threatening. Valid and reliable assessment is essential for effective pain management. The very nature of pain makes it impossible to measure objectively. There are different types of pain, and as caregivers, we need to diagnose the pain accurately in order that each patient gets the most effective treatment and continued evaluations, as needed. When caregivers decide on a treatment for pain, they are relying on the relatively objective VAS (Visual Analogue Scale.) According to recent studies most patients were dissatisfied with the pain treatment they had received. Approximately eighty percent of patients who present to emergency departments worldwide come because of pain.

Often the patient and the caregiver have different ideas about what pain is and how to treat it. Cultural differences, gender differences, even age differences may affect reactions of both the caretaker and the patient. There are many ways to treat pain, and various reasons for how people react to pain.

The present study is designed to measure the knowledge and attitudes of caregivers and in regard to the pain of their patients. An assessment of patient satisfaction to pain management will be also be performed.

Staff members working in wards involved with pain will be asked to fill out anonymous questionnaires concerning knowledge and attitudes toward pain. Patients will also be asked to fill out anonymous questionnaires in regard to their pain treatment. Informed consent will be requested. Responses will be collated and recorded. A future study is planned using a new pain protocol. The questionnaires will be repeated after the protocol has been in place for 12 months, at which time responses will be compared.

ELIGIBILITY:
Inclusion Criteria:

Staff from the Ziv Medical Center and patients

Exclusion Criteria:

Staff members that do not deal with pain treatment

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population includes patients in pain.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Improvement of pain treatment for the patient | A 6-month assessment will be performed

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel